CLINICAL TRIAL: NCT06643923
Title: Investigation of the Effects of Lumbopelvic Stabilization-based Physiotherapy and Rehabilitation Training on Lower Urinary Tract Symptoms in Children With Duchenne Muscular Dystrophy and Lower Urinary Tract Dysfunction
Brief Title: Effects of Lumbopelvic Stabilization-based Physiotherapy and Rehabilitation Training in Duchenne Muscular Dystrophy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Demet Öztürk, Research Assistant, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024232; Lokman hekim university (Other: Lokman hekim university)
Record Dates: First submitted 2024-10-07; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Duchenne Muscular Dystrophy (DMD); Lower Urinary Track Symptoms
Keywords: Duchenne muscular dystrophy; lower urinary tract symptoms; urotherapy; lumbopelvic exercise; physiotherapy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Lower Urinary Tract Symptoms | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Children and their families who have scored 8.5 or higher on the DVSS will be invited for further evaluation. Participants will be divided into two groups (Treatment and Active Control) using a 6-way block randomization method among the volunteer families.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Both groups of participants will receive the same urotherapy education from the same therapist (Demet Öztürk). Following the education, both groups will be instructed to implement the lifestyle changes taught during the urotherapy education for a period of eight weeks. In addition to the education, the treatment group will receive online, supervised exercise sessions based on lumbopelvic stabilization exercises, administered by the physiotherapist. The exercise program has been designed according to the FITTEA principle, which is one of the key principles in exercise prescription.
  Interventions: Other: Exercise; Behavioral: Urotherapy
- Active Control (Active Comparator): Approximately 1.5 hours of urotherapy training will be given and the patient will be asked to apply the lifestyle changes learned in this training for 8 weeks.
  Interventions: Behavioral: Urotherapy

INTERVENTIONS:
Other: Exercise — F (Frequency): 3 days per week, with a total of 24 sessions. I (Intensity): Low to moderate intensity exercises with progression, ensuring no fatigue is induced.
  T (Time): Each session will last 30 minutes, over a total period of 8 weeks.
  T (Type):
  Warm-up exercises Core stabilization exercises: Aimed at improving core stability. Cool-down exercises E (Enjoyment): Gamified exercises, with sessions conducted to music. A (Adherence): A follow-up system will be implemented, including reminder notes and regular sending of session links to ensure compliance.
  Arms: Treatment
Behavioral: Urotherapy — The urotherapy education program was developed by an expert physiotherapist and was piloted with the families of children with DMD (16 parents) prior to the study. Pre-test and post-test assessments demonstrated that the knowledge level of DMD families increased after the training. Additionally, results from the satisfaction survey indicated a high level of satisfaction among the families regarding the urotherapy education (Mean satisfaction score: 33.875/35.000, Minimum=28, Maximum=35). Therefore, it was deemed appropriate to deliver the same urotherapy presentation to the DMD families within the scope of this study. The training lasts approximately 1 hour and will be delivered to families via an online method. Each family will receive the education individually, and no group sessions will be conducted.

SUMMARY:
This study aims to examine the effectiveness of supervised lumbopelvic stabilization in relation to factors associated with lower urinary tract symptoms in children diagnosed with Duchenne Muscular Dystrophy (DMD) who have lower urinary tract dysfunction. Children aged between 8 and 12 years, at stages 1-4 according to the Vignos scale, and who have a score of 8.5 or higher on the Dysfunctional Voiding Symptom Score (DVSS), will be included in the study. Demographic information will be collected through a general assessment form, while lower urinary tract symptoms will be assessed using the DVSS, a researcher-developed evaluation form, and a three-day bladder diary. Bowel symptoms will be evaluated using the Rome IV criteria and a seven-day bowel diary. Physical performance will be assessed via the Timed Up and Go Test and Gower's Test, muscle strength using the microFET2 hand dynamometer, lumbar lordosis angle with a Bubble inclinometer, participation in daily living activities via the Barthel Index, and perceived well-being of both the child and the parent will be assessed using the Faces Rating Scale. Participants will be randomly assigned to two groups (Treatment and Active Control) using a block randomization method. In the Active Control group, children will receive only urotherapy education. In the Treatment group, children will receive supervised, online, lumbopelvic exercise-based physiotherapy and rehabilitation sessions, in addition to urotherapy, conducted by a physiotherapist. The sessions will last eight weeks, with a total of 24 sessions. At the end of the eight-week period, both groups will be re-evaluated using the same assessment methods. Intra-group and inter-group comparisons will be completed using appropriate analytical methods.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with DMD by a specialist physician,
* Having received a score of 8.5 or higher on the Voiding Disorders Symptom Score (VMSS),
* Being between the ages of 8-12,
* Continuing ambulation (Vignos Scale Stage 1-4),
* Volunteering to participate in the study by parents and reading and signing the informed consent form.

Exclusion Criteria:

* Having another neuromuscular disease diagnosed other than DMD and/or accompanying DMD,
* Having family and/or child having cooperation problems in completing the evaluations for any reason,
* Lack of internet infrastructure or technical infrastructure that may cause difficulty in continuing distance education/follow-up,
* Having difficulty in understanding and speaking the Turkish language.

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Duchenne muscular dystrophy is an X-linked recessive hereditary disease. For these reasons, women can only be carriers. Diagnosed individuals are only men.
Enrollment: 34 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Lower urinary tract symptoms assessment | 8 weeks
  Lower urinary tract symptoms will be assessed with the UIRS questionnaire. UIRS questions the frequency of lower urinary tract symptoms in the last month and measures the severity of lower urinary tract dysfunction. Akbal et al. stated that a score of 8.5 is the optimum threshold value and that this value can be used to determine whether there are functional voiding symptoms. This cut-off value will be used as the inclusion criterion in our study. In addition to the UIRS, a three-day bladder diary (voiding diary, frequency-volume chart) will be used to assess lower urinary tract symptoms. This diary allows recording bladder functions and facilitates follow-up by documenting them. In addition, it is a practical, repeatable, valid and reliable assessment method. Before the diaries are given, individuals will definitely be given training on how to fill out the diary and what to look for when filling out the diary.

SECONDARY OUTCOMES:
Bowel symptom assessment | 8 weeks
  Due to the close relationship between bladder and bowel function, both systems should be screened in routine evaluations. In our study, bowel symptoms will be evaluated with the Rome IV criteria and a 7-day bowel diary. A form including the Bristol Stool Scale is applied in the bowel diary evaluation. With this diary; information can be obtained on defecation frequency, defecation times, stool form, presence of pain during defecation, presence of fecal incontinence, times and severity of fecal incontinence.
  Rome IV criteria are listed below:
  2 or fewer defecations per week, maneuvering to postpone defecation, feeling of a large stool mass in the rectum, painful and difficult bowel movements, stool thick enough to block the toilet hole, and a history of fecal incontinence at least once a week. The presence of at least 2 of these criteria and their persistence for at least 3 months is considered constipation.
Physical performance assessment | 8 weeks
  Physical performance will be assessed with the Timed Up and Go Test. The Timed Up and Go Test provides information about the mobility and balance of individuals. It is a valid, practical and objective assessment method for the pediatric population. It is a functional test and evaluates the individual's ability to stand up from a chair independently, walk a distance of three meters, turn activities and sit down on a chair independently. The test will begin after the child is explained in detail and demonstrated by the physiotherapist. The physiotherapist will measure the test with a stopwatch and record it in seconds.
Muscle strength assessment | 8 weeks
  In our study, the proximal muscle groups in and around the trunk will be measured. These muscles include trunk flexors, trunk extensors, hip flexors and quadriceps femoris muscles.
  The Hoggan microFET2 (Hoggan Scientific, LLC, Salt Lake City UT, USA) device will be used in muscle strength measurement. The Hoggan hand-held dynamometer has been shown to be a valid and reliable technique for muscle strength assessment in muscle diseases.
  Two types of tests are used in the use of the Hoggan microFET2 device, which is a hand-held dynamometer type: "make" and "break". For the make test, the researcher applies resistance in a fixed position and the subject is asked to show maximum effort. For the break test, the researcher tries to apply more resistance than the maximum resistance shown by the subject, causing movement in the opposite direction of the joint. In our study, the "make" test will be used in order not to increase fatigue in children with DMD.
Lumbar lordosis angle assessment | 8 weeks
  Lumbar lordosis assessment will be performed while the person is standing without shoes, knees extended and feet hip-width apart. The person will be asked to fix their gaze on a single point at eye level and to keep their upper extremity freely near their hips. The person will be asked to stand comfortably while standing and if they voluntarily straighten up, the measurement will be repeated. In the lumbar lordosis measurement, 2 reference points will be marked and the Bubble inclinometer will be placed at these reference points and the measurement will be made from the sagittal plane. The first reference point is the lumbosacral segment and is S1-S2. The second reference point is the thoracolumbar segment and is at the T12-L1 level. The sum of the values measured from these two points gives the lumbar lordosis angle. The reference points will be marked with a pen that does not harm the skin.
Evaluation of participation in daily living activities | 8 weeks
  According to the recommendations of the International Classification of Functioning, Disability and Health (ICF), which is considered important by the World Health Organization, humans are biopsychosocial beings and should be evaluated in terms of psychosocial and participation as well as physical symptoms. Therefore, our study aimed to evaluate the participation and independence of the participants.
Perceived well-being assessment | 8 weeks
  Perceived well-being is different from physical parameters and is measured subjectively. The Facial Expression Scale will be used for the assessment of perceived well-being in the study. In addition, the perceived well-being assessment will be applied to both the parent and the child. The Facial Expression Scale is recommended for use in cases where the use of the visual analog scale and/or numerical scale is difficult and in children.
Physical performance assessment | 8 weeks
  Physical performance will be assessed with the Gowers Test. The Gowers is a timed performance test and is frequently used in individuals with DMD. For this test, the child will lie on his/her back on a mat spread on the floor. Then, the child will be asked to stand up as quickly as possible and come to an upright position. During the test, the physiotherapist will time the time it takes to stand up in.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Undecided